CLINICAL TRIAL: NCT07322991
Title: A Phase 1 Clinical Trial With an Open-label, Single-agent Repeated Dosing Followed by Combined Repeated Dosing Design to Evaluate the Drug-drug Interaction Between IY001 and IY002 in Healthy Adult Male Subjects.
Brief Title: Study to Evaluate the Drug-drug Interaction Between IY001 and IY002 in Healthy Adult Male Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IY-DDI2025
Record Dates: First submitted 2025-12-11; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-10

CONDITIONS: Healthy Adult Male
Keywords: Urology; Drug-Drug Interaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A (Experimental): IY001 -> IY001 + IY002
  Interventions: Drug: IY001(Finasteride); Drug: IY002(Tamsulosin)
- Part B (Experimental): IY002 -> IY001 + IY002
  Interventions: Drug: IY001(Finasteride); Drug: IY002(Tamsulosin)

INTERVENTIONS:
Drug: IY001(Finasteride) — Subjects will receive IY001 once daily for 3 days, followed by co-administration of IY001 and IY002 once daily for 5 days.
Drug: IY002(Tamsulosin) — Subjects will receive IY002 once daily for 5 days, followed by co-administration of IY001 and IY002 once daily for 3 days.

SUMMARY:
The purpose of this stud is to evaluate the drug-drug interaction between IY001 and IY002 in adult males.

DETAILED DESCRIPTION:
The study is an Open-label, Phase I, drug-drug interaction study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males aged between 19 and 55 years at screening.
* Body weight ≥ 50 kg and body mass index (BMI) between 18 and 30 kg/m² (BMI calculated as weight [kg] / height [m]²).
* No clinically significant congenital or chronic diseases, and no pathological signs or symptoms based on internal medicine examination (including EEG, ECG, chest or upper gastrointestinal endoscopy, or gastrointestinal radiographic examination, if necessary).
* Considered suitable for participation by the principal investigator (or delegated sub-investigator) based on diagnostic tests such as hematology, blood chemistry, serology, urinalysis, ECG, suicide risk assessment, and depression scale evaluation conducted in accordance with the characteristics of the investigational drugs.
* Able to provide written informed consent after receiving a detailed explanation of the clinical trial and voluntarily agreeing to participate and comply with study requirements during the trial period.
* Agree to use highly effective contraception* (excluding hormonal methods) and refrain from donating sperm from the first dose until at least 4 weeks after the last dose of the investigational drugs. This includes agreement that the subject or their partner will avoid pregnancy.

  *Highly effective contraception methods include: intrauterine device (IUD), bilateral tubal ligation, vasectomy of partner, or sexual abstinence. Methods such as periodic abstinence (calendar method, basal body temperature, ovulation method), withdrawal, use of spermicides alone, lactational amenorrhea, or simultaneous use of male and female condoms are not considered effective contraception.
* Agree not to donate blood from the first dose until at least 4 weeks after the last dose of the investigational drugs.

Exclusion Criteria:

* Use of drug-metabolizing enzyme inducers or inhibitors (e.g., barbiturates) within 30 days prior to the first dose, or use of such medications within 10 days prior to the first dose.
* Participation in a bioequivalence study or other clinical trial involving investigational drugs within 6 months prior to the first dose.
* Whole blood donation within 8 weeks, plasma donation within 2 weeks, or blood transfusion within 4 weeks prior to the first dose.
* History of gastrointestinal surgery that may affect drug absorption (excluding appendectomy and hernia surgery).
* Within 1 month prior to the first dose:

  * Average alcohol consumption exceeding 21 drinks per week (1 drink = 50 mL soju, 250 mL beer, or 30 mL spirits)
  * Smoking more than 20 cigarettes per day
* Any of the following conditions:

  * History of hypersensitivity (including angioedema) to the investigational drug or its components
  * Orthostatic hypotension
  * Severe hepatic impairment
  * Severe renal impairment
  * Currently taking PDE5 inhibitors
  * Currently taking CYP3A4 inhibitors
  * Currently taking antihypertensive drugs
  * Currently taking alpha-1 blockers
  * History of micturition syncope
  * Genetic disorders such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
  * Hypersensitivity or allergy to Sunset Yellow FCF (Yellow No. 5) contained in the drug
* History of clinically significant psychiatric disorders.
* Any other condition that the principal investigator (or delegated sub-investigator) deems makes the subject unsuitable for participation in this clinical trial.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study enrolls only male participants because the Investigational Product contain ingredients contraindicated for use in females.
Enrollment: 43 (Actual)
Dates: Start 2025-10-14 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Finasteride Area Under the Curve during the dosing interval at steady state (AUCτ,ss) | Measured at steady state after repeated dosing.(Day 8 compared to Day 3)
  The total drug exposure of finasteride over the dosing interval at steady state.
Finasteride Maximum Plasma Concentration at steady state (Cmax,ss) | Measured at steady state after repeated dosing.(Day 8 compared to Day 3)
  The peak plasma concentration of finasteride observed at steady state.
Tamsulosin Area Under the Curve during the dosing interval at steady state (AUCτ,ss) | Measured at steady state after repeated dosing.(Day 8 compared to Day 5)
  The total drug exposure of tamsulosin over the dosing interval at steady state.
Tamsulosin Maximum Plasma Concentration at steady state (Cmax,ss) | Measured at steady state after repeated dosing.(Day 8 compared to Day 5)
  The peak plasma concentration of tamsulosin observed at steady state.

SECONDARY OUTCOMES:
Finasteride Time to Maximum Plasma Concentration at steady state (Tmax,ss) | Days 3 and 8
  Time to reach the maximum plasma concentration of finasteride measured from plasma samples collected at pre-dose and multiple post-dose time points on Days 3 and 8.
Finasteride Elimination Half-Life at Steady State (t1/2,ss) | Days 3 and 8
  The elimination half-life of finasteride calculated using plasma concentrations from serial blood samples collected up to 24 hours post-dose on Days 3 and 8.
Finasteride Apparent Clearance at Steady State (CLss/F) | Days 3 and 8
  Apparent clearance of finasteride derived from plasma concentration-time data obtained from serial blood sampling on Days 3 and 8.
Finasteride Minimum Plasma Concentration at Steady State (Cmin,ss) | Days 1, 2, 7, and 8
  Minimum plasma concentration measured from pre-dose (0 hour) samples collected on Days 1, 2, 7, and 8.
Finasteride Average Plasma Concentration at Steady State (Cav,ss) | Days 3 and 8
  Average plasma concentration calculated over the dosing interval from serial samples collected on Days 3 and 8.
Finasteride Accumulation Ratio (R) | Days 3 and 8
  Ratio of plasma concentrations comparing steady state (Day 8) to earlier dosing period (Day 3).
Finasteride Peak-Trough Fluctuation (PTF) | Days 3 and 8
  Fluctuation between peak (Cmax) and trough (Cmin) plasma concentrations calculated from serial sampling on Days 3 and 8.
Tamsulosin Time to Maximum Plasma Concentration at Steady State (Tmax,ss) | Days 5 and 8
  Time to reach the maximum plasma concentration of tamsulosin measured from plasma samples collected at pre-dose and multiple post-dose time points on Days 5 and 8.
Tamsulosin Elimination Half-Life at Steady State (t1/2,ss) | Days 5 and 8
  Elimination half-life calculated from plasma concentrations obtained up to 24 hours post-dose on Days 5 and 8.
Tamsulosin Apparent Clearance at Steady State (CLss/F) | Days 5 and 8
  Apparent clearance derived from plasma concentration-time data on Days 5 and 8.
Tamsulosin Minimum Plasma Concentration at Steady State (Cmin,ss) | Days 1, 4, 7, and 8
  Minimum plasma concentration measured from pre-dose samples collected on Days 1, 4, 7, and 8.
Tamsulosin Average Plasma Concentration at Steady State (Cav,ss) | Days 5 and 8
  Average plasma concentration over dosing interval calculated from serial samples on Days 5 and 8.
Tamsulosin Accumulation Ratio (R) | Days 5 and 8
  Ratio of plasma concentrations comparing steady state (Day 8) to earlier dosing period (Day 5).
Tamsulosin Peak-Trough Fluctuation (PTF) | Days 5 and 8
  Fluctuation between peak (Cmax) and trough (Cmin) plasma concentrations from serial sampling on Days 5 and 8.

CONTACTS AND LOCATIONS:
Locations (1):
- H plus Yangji Hospital, Seoul, Seoul, South Korea